CLINICAL TRIAL: NCT04069078
Title: Prophylactic Use of Iv Hyoscine Butylbromide for Prevention of Bradycardia During Cesarean Section Under Spinal Anaesthesia. a Randomized Controlled Trial
Brief Title: Hyoscine Butylbromide for Prevention of Bradycardia During Cesarean Section
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Samy Abbas, associate professor of anesthesia, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: hyoscine
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-03

CONDITIONS: Bradycardia; Spinal Anesthetics Causing Adverse Effects in Therapeutic Use; Cesarean Section Complications
MeSH Terms: conditions — Bradycardia | interventions — Butylscopolammonium Bromide; Solutions; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hyoscine butylbromide (Active Comparator)
  Interventions: Drug: Hyoscine Butylbromide 20 Mg/mL Solution for Injection Ampoule
- Control (Placebo Comparator)
  Interventions: Other: Normal saline

INTERVENTIONS:
Drug: Hyoscine Butylbromide 20 Mg/mL Solution for Injection Ampoule — Patients will receive IV study solution which is hyoscine butylbromide 20 mg in 1 ml one minute after spinal anaesthesia
  Arms: Hyoscine butylbromide
Other: Normal saline — Patients will receive 1 ml of IV normal saline as a placebo one minute after spinal anesthesia
  Arms: Control

SUMMARY:
The aim of this study is to assess the efficacy of Iv hyoscine butylbromide in preventing Bradycardia during cesarean section under spinal anaesthesia with local anaesthetic and morphine.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status class I-II.
* Age: 18 Years to 40 Years.
* Women scheduled for elective Cesarean section under spinal anesthesia.
* indications for CS other than fetal or maternal pathology.

Exclusion Criteria:

* Height < 150 or > 180 cm
* Body mass index (BMI) >35 kg/m2
* Contraindication for central neuraxial block
* Refusal to undergo regional anesthesia
* Known allergy to any of the study drugs,
* Infection at the site of injection,
* Coagulopathy,
* Indication to general anesthesia
* Baseline bradycardia (heart rate < 60/min), or any cardiovascular disease
* Patients taking β-adrenergic blockers or any drugs that may alter normal response to study drugs.
* Arrhythmia such as atrial fibrillation, supraventricular tachycardia, heart block greater than first degree, left bundle branch block,
* Hypertension (systolic blood pressure more than 140 mm Hg or diastolic blood pressure more than 90 mm Hg), unstable angina or cardiomyopathy,
* Associated medical problem with pregnancy (as hypertension, diabetes mellitus, hepatic impairment or renal impairment)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 173 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2020-02-25 (Actual)

PRIMARY OUTCOMES:
Bradycardia | intraoperative
  number of participants who will develop heart rate below 50 BPM.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University hospital, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Abbas MS, Hassan SA, Abbas AM, Thabet AM, Thabet AM, Mahdy MM. Hemodynamic and antiemetic effects of prophylactic hyoscine butyl-bromide during cesarean section under spinal anesthesia: a randomized controlled trial. BMC Anesthesiol. 2022 Apr 21;22(1):112. doi: 10.1186/s12871-022-01659-9. PMID 35448942